CLINICAL TRIAL: NCT03347071
Title: Effects of a Yoga-Based Course in Preventing Disordered Eating in Female Collegiate Athletes: A Controlled Study
Brief Title: Effects of a Yoga-Based Course in Preventing Disordered Eating in Female Collegiate Athletes
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Give Back Yoga Foundation (Other)
Responsible Party: Principal Investigator, Catherine Cook-Cottone, Counseling, School, and Educational Psychology Associate Professor, Ph.D., University at Buffalo
Other Study IDs: EBTSA01
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2020-09

CONDITIONS: Disordered Eating Behaviors
Keywords: prevention; collegiate athletes; yoga
MeSH Terms: conditions — Disordered Eating Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prevention Course Group: The Prevention Course Group is composed of female student-athletes enrolled in the 7-week prevention course. The course occurs once a week (1 hour, 40 minute sessions) for a total of 7-weeks during the academic semester. Approximately 1 hour of each class session is lecture based, leaving 40 minutes for yoga practice administered by a certified yoga instructor. The course instructor is certified in Eat Breathe Thrive Program delivery. The course teaching assistant is certified in yoga instruction.
  Interventions: Behavioral: Prevention Course Group
- Control Group: The Control Group is composed of female student-athletes not enrolled in the 7-week prevention course. Female student-athletes in this group will not be enrolled in the course during the period of data collection, nor will they have previously completed the course.

INTERVENTIONS:
Behavioral: Prevention Course Group — The undergraduate prevention course is structured around Eat Breathe Thrive Program curriculum. The course aims to teach somatic practices, provide healthy tools for emotional regulation, allow for the creation of community-based networks of support, foster a sense of meaning and purpose through service activities, and practice these learned skills through yoga.
  Other Names: Eat Breathe Thrive Program
  Groups: Prevention Course Group

SUMMARY:
The purpose of the study is to evaluate effects of a 7-week undergraduate course, incorporating Eat Breathe Thrive program curriculum, offered to female student-athletes in order to increase positive body image, emotional regulation, interoceptive awareness, self-care skills, and intuitive eating. The undergraduate course is structured around the Eat Breathe Thrive program curriculum, which aims to: a) teach somatic practices that increase interoceptive awareness, b) provide healthy tools for emotional regulation, c) allow for the creation of community-based networks of support, and (d) foster a sense of meaning and purpose through service activities. In a non-randomized controlled trial, the investigators plan to examine whether this preventative undergraduate course is found effective in a female student-athlete population in preventing and decreasing eating disorder risk. The investigators also plan to examine whether the program is found effective in increasing protective factors, such as self-care behaviors, interoceptive awareness, intuitive eating, and emotional regulation skills.

DETAILED DESCRIPTION:
To the investigators' knowledge, there are no studies that incorporate yoga into eating disorder prevention intervention in a student-athlete population, indicating a gap in literature that the proposed study aims to address. In this study, a 7-week undergraduate course offered to female student-athletes, which incorporates Eat Breathe Thrive program curriculum, will be examined to evaluate preventative effects. The Eat Breathe Thrive program was selected by the course instructors to provide female student-athletes with mental health support, utilizing an interactive multisession format with a positive psychology orientation. Eat Breathe Thrive's curriculum focuses on the reduction of eating disorder risk by lesson plans centered around positive engagement with others and developing a strong relationship with self. This framework is based on the idea that individuals are able to sustain proper health, relationships, and overall well-being using the positive embodiment tools and psychoeducational information learned. The study aims to contribute to the eating disorder literature targeting female student-athletes by examining the effects of a prevention program delivered as part of an undergraduate course.

It is hypothesized that:

* Prevention course participants will show a decrease in disordered eating behaviors when compared to controls.
* Prevention course participants will show an increase in self-care behaviors compared to controls.
* Prevention course participants will show an increase in interoceptive awareness, intuitive eating, and emotional regulation when compared to controls.
* Prevention course participants will show a decrease in difficulties with emotional regulation and an increase in tolerance to distress when compared to controls.
* Prevention course participants will show better maintenance of wellbeing as well as better maintenance in decreased symptomatology as compared to compared to controls.

The study will employ self-report surveys to examine the preventative effects of participation in a 7-week course utilizing a longitudinal non-randomized control design with Division I female student-athletes in western New York. Participants will be current female student-athletes recruited within the university's athletic department. Experimental group participants will be recruited from their enrollment in the prevention course offered that incorporates the Eat Breathe Thrive curriculum. Since the prevention course has a capacity of 30 students per semester, data will be collected for four 7-week semesters to account for total sample size. The study will be recruiting from a total of 120 female student-athletes in the experimental group. Female student-athletes not enrolled in the prevention course will be recruited for control. Each semester, course enrollment numbers will be matched by recruiting research participants from the rest of the female student-athlete population at the university (those who are not enrolled in the course). Female student-athletes in the experimental and control groups will complete all study measures at the same time points throughout the study. This study is based on the need to provide female student-athletes with greater access to effective tools and strategies that support their well-being as well as to protect this high-risk population against the development of an eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a female undergraduate student-athletes at the university

Exclusion Criteria:

* There are no exclusion criteria not already covered within the criteria for inclusion stated

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are from the undergraduate student-athlete population at the university who are currently a member of one of the Division I sports teams. Specifically, female undergraduate student-athletes, ranging from ages 18-24.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Disordered Eating Behaviors | Change from Baseline in Eating Disorder Examination Questionnaire at 7 weeks
  Change in Eating Disorder Examination Questionnaire
Self-Care Behaviors | Change from Baseline in Mindful Self-Care Scale-Short at 7 weeks
  Change in Mindful Self-Care Scale-Short
Interoceptive Awareness | Change from Baseline in Multidimensional Assessment of Interoceptive Awareness at 7 weeks
  Change in Multidimensional Assessment of Interoceptive Awareness
Emotional Regulation | Change from Baseline in Difficulties in Emotion Regulation Scale at 7 weeks
  Change in Difficulties in Emotion Regulation Scale
Distress Tolerance | Change from Baseline in Distress Tolerance Scale and State-Trait Anxiety Inventory for Adults at 7 weeks
  Change in Distress Tolerance Scale and State-Trait Anxiety Inventory for Adults
Intuitive Eating | Change from Baseline in Intuitive Eating Scale in 7 weeks
  Change in Intuitive Eating Scale

SECONDARY OUTCOMES:
Disordered Eating Behaviors | Change from Baseline in Eating Disorder Examination Questionnaire at 19 weeks
  Change in Eating Disorder Examination Questionnaire
Self-Care Behaviors | Change from Baseline in Mindful Self-Care Scale-Short at 19 weeks
  Change in Mindful Self-Care Scale-Short
Emotional Regulation | Change from Baseline in Difficulties in Emotion Regulation Scale at 19 weeks
  Change in Difficulties in Emotion Regulation Scale
Distress Tolerance | Change from Baseline in Distress Tolerance Scale and State-Trait Anxiety Inventory for Adults at 19 weeks
  Change in Distress Tolerance Scale and State-Trait Anxiety Inventory for Adults

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cook-Cottone, PhD, Principal Investigator — Counseling, School, and Educational Psychology
Locations (1):
- Center for Excellence in Academic and Athletic Performance, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Curriculum offered in the prevention course is from the Eat Breathe Thrive Program — http://www.eatbreathethrive.org/